CLINICAL TRIAL: NCT03414593
Title: Prospective, Randomized, Single Blind Trial of Preemptive Analgesic Effects of Popliteal Sciatic Nerve Block in Patients With Bilateral Hallux Valgus Surgery
Brief Title: Preemptive Analgesic Effects of Popliteal Sciatic Nerve Block in Patients With Bilateral Hallux Valgus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hyuk Lee, clinical assistant professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017-0856
Record Dates: First submitted 2018-01-15; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Pain, Postoperative; Preemptive Peripheral Nerve Block; Acute Pain
Keywords: preemptive analgic effect; popliteal sciatic nerve block; Bilateral Hallux Valgus
MeSH Terms: conditions — Pain, Postoperative; Acute Pain

STUDY DESIGN:
Intervention Model Description: Patients who underwent surgery on both feet at the same time. One foot is performed before surgery and the other is performed after surgery.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoperative blocked leg: group preB (Experimental): ultrasound guided popliteal sciatic nerve block with 0.2% ropivacaine 20ml Before surgical incision
  Interventions: Drug: Ultrasound guided popliteal sciatic nerve block with 0.2% ropivcaine
- postoperative blocked leg: group postB (Active Comparator): ultrasound guided popliteal sciatic nerve block with 0.2% ropivacaine 20ml After surgical incision
  Interventions: Drug: Ultrasound guided popliteal sciatic nerve block with 0.2% ropivcaine

INTERVENTIONS:
Drug: Ultrasound guided popliteal sciatic nerve block with 0.2% ropivcaine — Ultrasound guided popliteal sciatic nerve block with 0.2% ropivacaine 20ml

SUMMARY:
The purpose of this study was to investigate the preemptive effect of ultrasound guided popliteal scistic nerve block on postoperative acute pain in patients with bilateral hallux valgus.

After induction of general anesthesia, the leg to be operated first is decided randomly. After the operation of one leg is completed, PSNB is performed on both legs with 0.2% Ropivacaine and surgery is started on the remaining legs.

When the surgery is over, check to see which foot pain begins first, how strong the pain is, and whether there are any side effects.

ELIGIBILITY:
Inclusion Criteria:

1. adults between the ages of 20 and 80
2. bilateral hallux valgus surgery on the same day
3. ASA class 1 or 2
4. Patients who have voluntarily agreed in writing to participate in the trial

Exclusion Criteria:

1. Patient with side effects on local anesthetics or steroids
2. Patient who are taboo of peripheral nerve block such as blood clotting disorder, infection, etc.
3. Patients with uncontrolled medical or psychiatric problem
4. Patient does not agree to participate in the study
5. Patients who are pregnant or lactating

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Analgesic duration of nerve block | at 0, 0.5, 1, 4, 8, 12 hours after operation. And AM 9 and PM 5 of POD (Post Operative Day) 1
  The difference of NRS during study time between group preB and group postB
  The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain. It is for adults and children 10 years old or older.
  0: No pain, 1-3: mild pain, 4-6: Moderate pain, 7-10: severe pain, 10: worst pain imaginable.

SECONDARY OUTCOMES:
Difference of analgesic consumption between both group | at 0, 0.5, 1, 4, 8, 12 hours after operation. And AM 9 and PM 5 of POD (Post Operative Day) 1
  The difference of usage of rescue analgesics during study time between group preB and group postB after the operation
side effect of popliteal sciatic nerve block | at 0, 0.5, 1, 4, 8, 12 hours after operation. And AM 9 and PM 5 of POD (Post Operative Day) 1
  any other sensation except pain

CONTACTS AND LOCATIONS:
Overall Officials: JongHyuk Lee, md, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea